CLINICAL TRIAL: NCT02915913
Title: Effects of High Intensity Interval- vs Resistance or Combined- Training for Improving Cognitive Function and Neurotrophic Factors in Overweight Adults (BrainFit Study): Factorial Randomised Controlled Trial
Brief Title: Effects of Exercise Training on Cognitive Function and Neurotrophic Factors in Overweight Adults
Acronym: BrainFit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Santo Tomas (Other)
Collaborators: Universidad del Rosario (Other); Universidad Nacional de Colombia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 2016-09-22
Record Dates: First submitted 2016-09-22; First posted 2016-09-27 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Cognitive Function; Motor Activity; Obesity
MeSH Terms: conditions — Motor Activity; Obesity | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- High Intensity Interval (Experimental): One session for 30-60 minutes of high intensity aerobic exercise
  Interventions: Behavioral: Experimental: High Intensity Interval
- Resistance training (Experimental): One session for 30-60 minutes of resistance exercise
  Interventions: Behavioral: Resistance training
- Plus: High Intensity Interval + Resistance Training (Experimental): One session for 30-60 minutes of high intensity aerobic exercise and resistance exercise
  Interventions: Behavioral: Plus: High Intensity Interval + Resistance Training
- Non-exercise (Placebo Comparator): Non-exercise
  Interventions: Other: Non-exercise

INTERVENTIONS:
Behavioral: Experimental: High Intensity Interval — Walking on a treadmill 4min at 80-90% peak heart rate and recovery 4 min at 65% peak heart rate until expenditure of 500 kcal
  Arms: High Intensity Interval
Behavioral: Resistance training — Completing a resistance circuit (including upper and lower muscle groups) as many times as needed according to subject weight until expenditure of 500 kcal
  Arms: Resistance training
Behavioral: Plus: High Intensity Interval + Resistance Training — Walking on a treadmill as intervention 1 until 50% the energy expenditure prescribed is reached, then completing a resistance circuit until 100% energy expenditure is reached
  Arms: Plus: High Intensity Interval + Resistance Training
Other: Non-exercise — This group will receive the usual clinical care according to the consensus recommendations of the national goals for cardiovascular health promotion and disease reduction of the American Heart Association and Colombian guidelines COLDEPORTES.
  Arms: Non-exercise

SUMMARY:
The BrainFit Study aims to examine acute effects of High Intensity Interval- vs Resistance or Combined program has benefits on Cognitive Function as well as on secretion and regulation of neurotrophic factors or neurotrophins in a cohort of sedentary, overweight adults (aged 18-30 years) from Bogota, Colombia.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Interested in improving health and fitness.
* Central obesity: waist circumference ≥90cm
* Body mass index ≥ 26 kg/m(2)

Exclusion Criteria:

* Systemic infections.
* Weight loss or gain of >10% of body weight in the past 6 months for any reason.
* Currently taking medication that suppresses or stimulates appetite.
* Uncontrolled hypertension: systolic blood pressure 160 mm Hg or diastolic blood pressure 95 mm Hg on treatment.
* Gastrointestinal disease, including self-reported chronic hepatitis or cirrhosis, any episode of alcoholic hepatitis or alcoholic pancreatitis within past year, inflammatory bowel disease requiring treatment in the past year, recent or significant abdominal surgery (e.g., gastrectomy).
* Asthma.
* Diagnosed diabetes (type 1 or 2), fasting impaired glucose tolerance (blood glucose 118 mg/dL), or use of any anti-diabetic medications.
* Currently taking antidepressant, steroid, or thyroid medication, unless dosage is stable (no change for 6 months).
* Any active use of illegal or illicit drugs.
* Current exerciser (>30 min organized exercise per week).
* Indication of unsuitability of current health for exercise protocol (PARQ).

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Brain-derived neurotrophic factor | Baseline and 60 minutes immediately after the interventions ends
  Measurement of serum Brain-derived neurotropic factor true blood samples.

SECONDARY OUTCOMES:
Change from Baseline in Neurotrophin-3 | Baseline and 60 minutes immediately after the interventions ends
Change from Baseline in Neurotrophin-4 | Baseline and 60 minutes immediately after the interventions ends
Change from Baseline change in Cognitive Function | Baseline and 60 minutes immediately after the interventions ends
  Cognitive Performance Test (BPT) computerized cognitive assessment battery developed by Lumos Labs, Inc.

CONTACTS AND LOCATIONS:
Overall Officials: Robinson Ramírez-Vélez, Ph.D, Study Director — Universidad del Rosario
Locations (1):
- Robinson Ramírez-Vélez, Bogota, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dominguez-Sanchez MA, Bustos-Cruz RH, Velasco-Orjuela GP, Quintero AP, Tordecilla-Sanders A, Correa-Bautista JE, Triana-Reina HR, Garcia-Hermoso A, Gonzalez-Ruiz K, Pena-Guzman CA, Hernandez E, Pena-Ibagon JC, Tellez-T LA, Izquierdo M, Ramirez-Velez R. Acute Effects of High Intensity, Resistance, or Combined Protocol on the Increase of Level of Neurotrophic Factors in Physically Inactive Overweight Adults: The BrainFit Study. Front Physiol. 2018 Jun 27;9:741. doi: 10.3389/fphys.2018.00741. eCollection 2018. PMID 29997519